CLINICAL TRIAL: NCT00477425
Title: Evaluation of Corrected QT Interval From Clinical Studies Conducted With Bevacizumab
Brief Title: A Study to Evaluate Corrected QT Interval From Clinical Studies Conducted With Bevacizumab
Status: Withdrawn | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Other Study IDs: AVF4223g
Record Dates: First submitted 2007-05-21; First posted 2007-05-23 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Carcinoma
Keywords: Avastin
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a supplemental study designed to evaluate the effect of bevacizumab on QTc interval in cancer patients. Patients who have consented to participate in selected randomized controlled bevacizumab clinical trials will be invited to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Enrollment in one of a list of certain randomized, controlled bevacizumab trials

Exclusion Criteria:

* Implantable pacemaker or automatic implantable cardioverter defibrillator (AICD)
* Congenital long QT syndrome
* Family history of long QT syndrome
* Clinically significant bradycardia (defined as < 50 beats/minute)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Huang, M.D., Study Director — Genentech, Inc.